CLINICAL TRIAL: NCT02785549
Title: Multicentre Controlled, Randomized Clinical Trial to Compare the Efficacy and Safety of Ambulatory Treatment of Mild Acute Diverticulitis Without Antibiotics With the Standard Treatment With Antibiotics
Brief Title: Randomized Clinical Trial to Compare the Treatment of Mild Acute Diverticulitis With or Without Antibiotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Neus Ruiz-Edo, MD, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIR-DISA-2016; 2016-001596-75 (EudraCT Number)
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Acute Diverticulitis
Keywords: Acute diverticulitis; Antibiotic; Outpatient treatment
MeSH Terms: interventions — Ibuprofen; Acetaminophen; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Symptomatic treatment with NSAID (Experimental): 1 g/8 h acetaminophen alternating with 600 mg/8 h ibuprofen
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen
- Antibiotic+symptomatic treatment with NSAID (Active Comparator): 875/125mg /8h amoxicillin/clavulanic acid and symptomatic treatment with 1 g/8 h acetaminophen alternating with 600 mg/8 h ibuprofen
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen; Drug: Amoxicillin/clavulanic acid

INTERVENTIONS:
Drug: Ibuprofen — 600 mg/8hours
Drug: Acetaminophen — 1 g/8 hours
  Other Names: Paracetamol
Drug: Amoxicillin/clavulanic acid — 875mg/125mg/8 hours
  Arms: Antibiotic+symptomatic treatment with NSAID

SUMMARY:
Patients with mild acute diverticulitis (modified Neff 0 grade), following the inclusion criteria and giving informed consent, will be included in the study protocol and will be randomly assigned to one of the treatment arms: symptomatic treatment with NSAID plus antibiotic vs symptomatic treatment with NSAID only. They will be followed-up at 48 hours, 7 days, 30 days and 3 months from the onset of the episode.

DETAILED DESCRIPTION:
In the last years, traditional pathologic mechanisms of acute diverticulitis are being questioned and replaced by more scientifically grounded hypotheses that strongly postulate an inflammatory origin. Local pro-inflammatory cytokines, microbiota shifts, disturbed neurological intestinal signalling due to alterations in colonic neuropeptides and abnormal colonic motility are all being proposed as potential etiologic factors. Recent publications, therefore, call into question the benefits of antibiotic treatment or episodes of acute diverticulitis, especially for mild episodes. Furthermore, recent international guidelines endorse this stance in their recommendations. Moreover, recent studies provide evidence regarding the security of treating patients with mild acute diverticulitis as outpatients.

The investigators think that outpatient treatment without antibiotic for mild acute diverticulitis is not-inferior to traditional treatment with antibiotic, measuring the efficacy with readmission ratio. For this reason we have designed a multicentric, randomised, prospective study.

All patients seen in the emergency department with clinical signs of acute diverticulitis (left iliac fossa abdominal pain, peritoneal irritation signs and/or leucocytosis) will undergo an abdominal computed tomography to confirm the diagnosis and grade the disease according to severity using the modified Neff (mNeff) classification. Those with mild acute diverticulitis (grade 0), following the inclusion criteria and giving informed consent, will be included in the study protocol and will be randomly assigned to one of the treatment arms: symptomatic treatment with NSAID plus antibiotic vs symptomatic treatment with NSAID only. They will be followed-up at 48 hours, 7 days, 30 days and 3 months from the onset of the episode.

Primary goal is to determine if, in mild acute diverticulitis, the treatment without antibiotic is not-inferior to the traditional treatment with antibiotic considering readmission ratio.

Secondary goals include the analysis of the differences between groups, in case there are, in relation to number and reason for reconsultation, reason for readmission (bad symptoms control, radiologic progression, analysis worsening), pain control (analogic visual scale), recuperation after the acute episode, complication rate and their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient's written informed consent. Adequate cognitive capacity.
* Adequate family support
* No acute diverticulitis episode in the last 3 months
* mNeff 0 acute diverticulitis (abdominal computed tomography scan)
* No antibiotic treatment in the last 2 weeks
* Immunocompetence*
* No significant comorbidities**
* Good oral tolerance
* Good symptom control
* Maximum one of the following SIRS criteria (* T>38 ºC or <36ºC, L>12,000 or <4000/uL, HR>90 bpm, RR<20 rpm) or CRP>15 mg/dL

Exclusion Criteria:

* Women in pregnancy or breastfeeding
* Age <18 years or > 80 years.
* Absence of the patient's written informed consent. Inadequate cognitive capacity.
* Inadequate family support
* Acute diverticulitis episode in the last 3 months
* Moderate acute diverticulitis (mNeff grade I or upper)
* Antibiotic treatment in the last 2 weeks
* Inflammatory bowel disease
* Immunodepression*
* Presence of significant comorbidities**
* Bad oral tolerance
* Poor symptom control
* More than one of the following SIRS criteria (* T>38 ºC or <36ºC, L>12,000 or <4000/uL, HR>90 bpm, RR<20 rpm) or CRP>15 mg/dL

(*) Immunocompetence is the absence and immunodepression is the presence of any of the following: active neoplastic disease/hematologic malignancy/HIV with low CD4+ count/long-term corticosteroid treatment/immunosuppressant therapy/transplant/splenectomy/genetic immunodeficiency.

(**) We consider significant comorbidities any of the following: poorly controlled diabetes mellitus (HbA1>7mg/dl), cardiologic event in the last 3 months, decompensation of hepatopathy in the last 3 months, renal chronic insufficiency in dialysis programme.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2016-11; Primary Completion 2020-01-12 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Readmission ratio | 3 months
  Primary outcome is to determine if, in mild acute diverticulitis, the treatment without antibiotic is not-inferior to the traditional treatment with antibiotic considering readmission ratio.

SECONDARY OUTCOMES:
Reconsultation ratio | 3 months
  The analysis of the differences between groups, in case there are, in relation to number and reason for reconsultation
Reason for reconsultation | 3 months
  The analysis of the differences between groups, in case there are, in relation to number and reason for reconsultation
Reason for readmission | 3 months
  The analysis of the differences between groups, in case there are, in relation to reason for readmission (bad symptoms control, radiologic progression, analysis worsening)
Pain control | 48 hours, 7 days, 1 month, 3 months
  The analysis of the differences between groups, in case there are, in relation to pain control (analogic visual scale), during follow-up.
Complications | 3 months
  Description of the complications in both groups (perforation, abscess) and its treatment (percutaneous drainage, emergency surgery, broad spectrum antibiotics)

CONTACTS AND LOCATIONS:
Overall Officials: Neus Ruiz, MD, Principal Investigator — Corporacion Parc Tauli; Laura Mora, MD PhD, Principal Investigator — Corporacion Parc Tauli
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Strate LL, Modi R, Cohen E, Spiegel BM. Diverticular disease as a chronic illness: evolving epidemiologic and clinical insights. Am J Gastroenterol. 2012 Oct;107(10):1486-93. doi: 10.1038/ajg.2012.194. Epub 2012 Jul 10. PMID 22777341
- [Background] Daniels L, Budding AE, de Korte N, Eck A, Bogaards JA, Stockmann HB, Consten EC, Savelkoul PH, Boermeester MA. Fecal microbiome analysis as a diagnostic test for diverticulitis. Eur J Clin Microbiol Infect Dis. 2014 Nov;33(11):1927-36. doi: 10.1007/s10096-014-2162-3. Epub 2014 Jun 4. PMID 24894339
- [Background] Espin F, Rofes L, Ortega O, Clave P, Gallego D. Nitrergic neuro-muscular transmission is up-regulated in patients with diverticulosis. Neurogastroenterol Motil. 2014 Oct;26(10):1458-68. doi: 10.1111/nmo.12407. Epub 2014 Aug 11. PMID 25109425
- [Background] Humes DJ, Simpson J, Smith J, Sutton P, Zaitoun A, Bush D, Bennett A, Scholefield JH, Spiller RC. Visceral hypersensitivity in symptomatic diverticular disease and the role of neuropeptides and low grade inflammation. Neurogastroenterol Motil. 2012 Apr;24(4):318-e163. doi: 10.1111/j.1365-2982.2011.01863.x. Epub 2012 Jan 25. PMID 22276853
- [Background] Chabok A, Pahlman L, Hjern F, Haapaniemi S, Smedh K; AVOD Study Group. Randomized clinical trial of antibiotics in acute uncomplicated diverticulitis. Br J Surg. 2012 Apr;99(4):532-9. doi: 10.1002/bjs.8688. Epub 2012 Jan 30. PMID 22290281
- [Background] Isacson D, Thorisson A, Andreasson K, Nikberg M, Smedh K, Chabok A. Erratum to: Outpatient, non-antibiotic management in acute uncomplicated diverticulitis: a prospective study. Int J Colorectal Dis. 2015 Sep;30(9):1235. doi: 10.1007/s00384-015-2284-9. No abstract available. PMID 26084881
- [Background] Estrada Ferrer O, Ruiz Edo N, Hidalgo Grau LA, Abadal Prades M, Del Bas Rubia M, Garcia Torralbo EM, Heredia Budo A, Sunol Sala X. Selective non-antibiotic treatment in sigmoid diverticulitis: is it time to change the traditional approach? Tech Coloproctol. 2016 May;20(5):309-315. doi: 10.1007/s10151-016-1464-0. Epub 2016 Apr 6. PMID 27053254
- [Background] Brochmann ND, Schultz JK, Jakobsen GS, Oresland T. Management of acute uncomplicated diverticulitis without antibiotics: a single-centre cohort study. Colorectal Dis. 2016 Nov;18(11):1101-1107. doi: 10.1111/codi.13355. PMID 27089051
- [Background] Unlu C, de Korte N, Daniels L, Consten EC, Cuesta MA, Gerhards MF, van Geloven AA, van der Zaag ES, van der Hoeven JA, Klicks R, Cense HA, Roumen RM, Eijsbouts QA, Lange JF, Fockens P, de Borgie CA, Bemelman WA, Reitsma JB, Stockmann HB, Vrouenraets BC, Boermeester MA; Dutch Diverticular Disease 3D Collaborative Study Group. A multicenter randomized clinical trial investigating the cost-effectiveness of treatment strategies with or without antibiotics for uncomplicated acute diverticulitis (DIABOLO trial). BMC Surg. 2010 Jul 20;10:23. doi: 10.1186/1471-2482-10-23. PMID 20646266
- [Background] Andersen JC, Bundgaard L, Elbrond H, Laurberg S, Walker LR, Stovring J; Danish Surgical Society. Danish national guidelines for treatment of diverticular disease. Dan Med J. 2012 May;59(5):C4453. PMID 22549495
- [Background] Andeweg CS, Mulder IM, Felt-Bersma RJ, Verbon A, van der Wilt GJ, van Goor H, Lange JF, Stoker J, Boermeester MA, Bleichrodt RP; Netherlands Society of Surgery; Working group from Netherlands Societies of Internal Medicine, Gastroenterologists, Radiology, Health echnology Assessment and Dieticians. Guidelines of diagnostics and treatment of acute left-sided colonic diverticulitis. Dig Surg. 2013;30(4-6):278-92. doi: 10.1159/000354035. Epub 2013 Aug 20. PMID 23969324
- [Background] Cuomo R, Barbara G, Pace F, Annese V, Bassotti G, Binda GA, Casetti T, Colecchia A, Festi D, Fiocca R, Laghi A, Maconi G, Nascimbeni R, Scarpignato C, Villanacci V, Annibale B. Italian consensus conference for colonic diverticulosis and diverticular disease. United European Gastroenterol J. 2014 Oct;2(5):413-42. doi: 10.1177/2050640614547068. PMID 25360320
- [Background] Kruis W, Germer CT, Leifeld L; German Society for Gastroenterology, Digestive and Metabolic Diseases and The German Society for General and Visceral Surgery. Diverticular disease: guidelines of the german society for gastroenterology, digestive and metabolic diseases and the german society for general and visceral surgery. Digestion. 2014;90(3):190-207. doi: 10.1159/000367625. Epub 2014 Nov 19. PMID 25413249
- [Background] Mora Lopez L, Serra Pla S, Serra-Aracil X, Ballesteros E, Navarro S. Application of a modified Neff classification to patients with uncomplicated diverticulitis. Colorectal Dis. 2013 Nov;15(11):1442-7. doi: 10.1111/codi.12449. PMID 24192258
- [Background] Alonso S, Pera M, Pares D, Pascual M, Gil MJ, Courtier R, Grande L. Outpatient treatment of patients with uncomplicated acute diverticulitis. Colorectal Dis. 2010 Oct;12(10 Online):e278-82. doi: 10.1111/j.1463-1318.2009.02122.x. PMID 19906059
- [Background] Biondo S, Golda T, Kreisler E, Espin E, Vallribera F, Oteiza F, Codina-Cazador A, Pujadas M, Flor B. Outpatient versus hospitalization management for uncomplicated diverticulitis: a prospective, multicenter randomized clinical trial (DIVER Trial). Ann Surg. 2014 Jan;259(1):38-44. doi: 10.1097/SLA.0b013e3182965a11. PMID 23732265
- [Background] Gargallo Puyuelo CJ, Sopena F, Lanas Arbeloa A. Colonic diverticular disease. Treatment and prevention. Gastroenterol Hepatol. 2015 Dec;38(10):590-9. doi: 10.1016/j.gastrohep.2015.03.010. Epub 2015 May 12. PMID 25979437
- [Background] Makela JT, Klintrup K, Rautio T. The role of low CRP values in the prediction of the development of acute diverticulitis. Int J Colorectal Dis. 2016 Jan;31(1):23-7. doi: 10.1007/s00384-015-2410-8. Epub 2015 Oct 31. PMID 26519151
- [Background] Makela JT, Klintrup K, Takala H, Rautio T. The role of C-reactive protein in prediction of the severity of acute diverticulitis in an emergency unit. Scand J Gastroenterol. 2015 May;50(5):536-41. doi: 10.3109/00365521.2014.999350. Epub 2015 Feb 9. PMID 25665622
- [Derived] Mora-Lopez L, Ruiz-Edo N, Estrada-Ferrer O, Pinana-Campon ML, Labro-Ciurans M, Escuder-Perez J, Sales-Mallafre R, Rebasa-Cladera P, Navarro-Soto S, Serra-Aracil X; DINAMO-study Group. Efficacy and Safety of Nonantibiotic Outpatient Treatment in Mild Acute Diverticulitis (DINAMO-study): A Multicentre, Randomised, Open-label, Noninferiority Trial. Ann Surg. 2021 Nov 1;274(5):e435-e442. doi: 10.1097/SLA.0000000000005031. PMID 34183510
- [Derived] Mora Lopez L, Ruiz-Edo N, Serra Pla S, Pallisera Llovera A, Navarro Soto S, Serra-Aracil X; Diverticulitis Study Group. Multicentre, controlled, randomized clinical trial to compare the efficacy and safety of ambulatory treatment of mild acute diverticulitis without antibiotics with the standard treatment with antibiotics. Int J Colorectal Dis. 2017 Oct;32(10):1509-1516. doi: 10.1007/s00384-017-2879-4. Epub 2017 Aug 14. PMID 28808771